CLINICAL TRIAL: NCT05966194
Title: A Randomized Placebo-Controlled Trial of Two Schedules of RRx-001 for the Attenuation of Severe Oral Mucositis in Patients Receiving Concomitant Chemoradiation for the Treatment of Locally Advanced Squamous Cell Carcinoma of the Oral Cavity or Oropharynx
Brief Title: RRx-001 for Reducing Oral Mucositis in Patients Receiving Chemotherapy and Radiation for Head and Neck Cancer
Acronym: KEVLARx
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-01
Record Dates: First submitted 2023-07-21; First posted 2023-07-28 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Oral Mucositis
Keywords: Head and Neck Cancer; Neck cancer; Oral cancer; Mucositis; Squamous cell carcinoma (SCC); HPV; Oropharynx; Oral cavity; IMRT
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms; Mouth Neoplasms; Mucositis; Carcinoma, Squamous Cell | interventions — RRx-001; Radiotherapy, Intensity-Modulated; Cisplatin; Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RRx-001 Pre-Treatment (8mg RRx-001) + Chemoradiation Therapy (CRT) (Experimental): Pretreatment consists of 8 mg RRx-001 given twice weekly during the 2 weeks prior to the start of CRT (4 doses total) followed by the CRT treatment period
  Interventions: Drug: RRx-001; Radiation: Intensity Modulated Radiation Therapy (IMRT); Drug: Cisplatin for injection 100 mg/m2
- RRx-001 Pre-Treatment (4mg RRx-001) + Chemoradiation Therapy (CRT) (Experimental): Pretreatment consists of 4 mg RRx-001 given twice weekly during the 2 weeks prior to the start of CRT (4 doses total) followed by the CRT treatment period.
  Interventions: Drug: RRx-001; Radiation: Intensity Modulated Radiation Therapy (IMRT); Drug: Cisplatin for injection 100 mg/m2
- Placebo Pre-Treatment + Chemoradiation Therapy (CRT) (Placebo Comparator): No doses of RRx-001 will be administered. Patients assigned to this arm will receive placebo twice weekly during the 2 weeks prior to the start of CRT followed by the CRT treatment period.
  Interventions: Radiation: Intensity Modulated Radiation Therapy (IMRT); Drug: Cisplatin for injection 100 mg/m2

INTERVENTIONS:
Drug: RRx-001 — RRx-001 for injection (4 mg or 8 mg)
  Arms: RRx-001 Pre-Treatment (4mg RRx-001) + Chemoradiation Therapy (CRT); RRx-001 Pre-Treatment (8mg RRx-001) + Chemoradiation Therapy (CRT)
Radiation: Intensity Modulated Radiation Therapy (IMRT) — Intensity Modulated Radiation Therapy of up to 72 Gy
Drug: Cisplatin for injection 100 mg/m2 — Cisplatin for injection 100 mg/m2

SUMMARY:
The purpose of this study is to determine if RRx-001, which is added on to the cisplatin and radiation treatment, reduces the incidence of severe oral mucositis in patients with head and neck cancers. All patients in this study will receive 7 weeks of standard of care radiation therapy given with the chemotherapy agent, cisplatin. Patients will receive RRx-001 or placebo before start of standard of care treatment.

DETAILED DESCRIPTION:
The standard treatment for head and neck cancer currently includes a chemotherapy drug called cisplatin that is given by intravenous (IV) infusion and radiation, which is delivered from a machine that precisely targets the tumor. One common and unfortunate side effect of treatment with cisplatin and radiation is oral mucositis, which refers to irritation of the lining of the mouth. Oral mucositis is a serious problem 1) because the open mouth sores from oral mucositis may lead to severe pain, nutritional problems and dehydration from an inability to eat and drink, an increased risk of infection from bacteria and fungus and delay or discontinuation of treatment and 2) because there is only one approved therapy to treat or prevent it.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed diagnosis of squamous cell carcinoma (SCC) of the oral cavity or oropharynx Note: Patients with primary cancers that are presumed to be of oropharyngeal origin may be included if they meet radiation field dosing criteria as specified in Inclusion Criterion #2 below. Unknown primaries which are HPV+ are acceptable. HPV determination must be made for all patients.
2. Radiation Treatment planned to receive standard IMRT with daily fractions of 2.0 to 2.2 Gy for a total cumulative dose of 60-72 Gy in conjunction with definitive or adjuvant chemotherapy. Planned radiation treatment fields must include at least two oral sites (soft palate, floor of mouth, buccal mucosa, tongue) that are each planned to receive a total of > 55 Gy. Patients who have had prior surgery are eligible, provided they have fully recovered from surgery, and patients who may have surgery in the future are eligible.
3. ECOG performance status ≤ 2.
4. Participants must have adequate organ and marrow function as defined below:

   • Absolute neutrophil count (ANC) ≥ 1,500 / mm3 2. Platelets ≥ 75,000 / mm3 3. Hemoglobin ≥ 9.0 g/dL
5. Adequate renal and liver function as indicated by:

   • Serum creatinine acceptable for treatment with cisplatin per institutional guidelines) 2. Total bilirubin ≤ 1.5 x upper-normal limit (ULN) 3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3.0 x ULN 4. Alkaline phosphatase ≤ 2.5 x ULN
6. Human papilloma virus (HPV) status in tumor must be documented using tumor immunohistochemistry for HPV-p16 or other accepted test (such as such as in situ hybridization) for patients with cancers of the oropharynx (Rooper et al, 2016, Martens 2017). HPV status at baseline optional for oral cavity tumors.
7. Age 18 years or older
8. Patient must consent to the access, review, and analysis of previous medical and cancer history, including imaging data, by the sponsor or a third party nominated by the sponsor.
9. Ability and willingness to understand and sign a written informed consent document.
10. Women of childbearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy.

    Note: A woman of child-bearing potential is any female (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
    * Has not undergone a hysterectomy or bilateral oophorectomy; or
    * Has not been postmenopausal for at least 12 consecutive months
11. Adequate visual access to permit examination of the following oral cavity sites: lips, buccal mucosa, floor of mouth, ventral and lateral tongue, and soft palate.

Exclusion Criteria:

1. Prior radiotherapy to the head and neck region.
2. Prior induction chemotherapy.
3. Tumors of the lips, salivary gland, nasopharynx, hypopharynx, or larynx.
4. Patients with simultaneous primaries
5. Stage IV, M1 (distant metastasis)
6. Prior or current use of approved or investigational anticancer agent other than those provided in this study.
7. Grade 3 or 4 dysphagia or odynophagia (National Cancer Institute Common Toxicity Criteria, version 5.0) or inability to eat a normal (solid) diet
8. Requirement at baseline for parenteral or gastrointestinal tube-delivered nutrition for any reason or prophylactic insertion of gastrostomy tube with dependency on tube feeding at baseline.
9. Malignant tumors other than squamous cell carcinoma of the head and neck within last 5 years, unless treated definitively and with low risk of recurrence in the judgment of the treating investigator.
10. Active infectious disease excluding oral candidiasis.
11. Presence of oral mucositis (WHO Score ≥ Grade 1) or other oral mucosal ulceration at baseline.
12. Untreated active oral or dental infection
13. Known history of human immunodeficiency virus or active hepatitis B or C.
14. Any significant medical diseases or conditions, as assessed by the investigators and sponsor that would substantially increase the medical risks of participating in this study (e.g, immunosuppression, uncontrolled diabetes, NYHA II-IV congestive heart failure, myocardial infarction within 6 months of study, severe chronic pulmonary disease or active uncontrolled infection, uncontrolled or clinically relevant pulmonary edema)
15. Use of the following within 48 hours of enrollment and duration of Oral Mucositis follow up: vitamin B12 (cobalamin) or synthetic vitamin B12, cyanocobalamin, or the vitamin B12 precursor, cobinamide, or any supplement or multivitamin with vitamin B12 or vitamin E in it since both vitamin B12 and vitamin E interact negatively with RRx-001.
16. Use of prebiotics and probiotics
17. Pregnant or nursing.
18. Known allergies or intolerance to cisplatin or other platinum-containing compounds.
19. Sjogren syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Severe Oral Mucositis (SOM) through Intensity-modulated radiation therapy (IMRT) | Estimated up to 18 Months
  The incidence of SOM defined as the proportion of patients with any WHO Grade >= 3 (severe to life threatening) oral mucositis during the observation period from the start of CRT through IMRT

SECONDARY OUTCOMES:
Duration of Severe Oral Mucositis (SOM) through Intensity-modulated radiation therapy (IMRT) | Estimated up to 18 Months
  Duration of SOM (through the last day of radiation therapy, DoSOM). Its principal analysis employs the probability of being in response (PBIR), an intuitive concept based on the realization that the duration of response which is quantified as the area under the curve delimited by the duration of exposure (x axis) and the response probability (y axis).
Duration of Severe Oral Mucositis (SOM) through 60 Gy | Estimated up to 18 Months
  Duration of SOM (through 60 Gy, DoSOM) is compared between RRx-001 arms and Placebo using a two-sided log-rank test.
Time to onset of Sever Oral Mucositis (ttSOM) | Estimated up to 18 Months
  Time onset to SOM (ttSOM) is defined as the time interval measured from the start of the observation period to the first time SOM is observed.
Incidence and severity of dysphagia | Estimated up to 18 Months
  Incidence and severity of dysphagia will be analyzed similarly to the primary efficacy endpoint.
Cumulative radiation dose to onset of SOM | Estimated up to 18 Months
  Cumulative radiation dose to onset of SOM is compared between RRx-001 arms and placebo
Incidence of grade 4 oral mucositis | Estimated up to 18 Months
  Incidence of grade 4 oral mucositis through 60 Gy
Narcotic use through resolution of SOM | Estimated up to 18 Months
  Narcotic use through resolution of SOM will be analyzed similarly to the cumulative radiation dose
Incidence of Severe Oral Mucositis through 60 Gy of the Radiation Treatment Plan | Estimated up to 18 Months
  incidence of SOM defined as the proportion of patients with any WHO Grade >= 3 (severe to life threatening) oral mucositis during the observation period from the start of CRT through 60 Gy
Progression free survival (PFS) | Estimated up to 24 Months
  Progression free survival (PFS)
Degree of Xerostomia | Estimated up to 24 Months
  Degree of Xerostomia as analyzed by validated Xerostomia questionnaire 'XQ'
Xerostomia duration | Estimated up to 24 Months
  Xerostomia duration as analyzed by validated Xerostomia questionnaire 'XQ'
Time to onset of dysphagia | Estimated up to 24 Months
  Time to onset of dysphagia
Duration of dysphagia | Estimated up to 24 Months
  Duration of dysphagia

CONTACTS AND LOCATIONS:
Overall Officials: Meaghan Stirn, Study Director — EpicentRx, Inc.
Locations (14):
- United States (14):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Miami Cancer Institute, Miami, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Parkview Cancer Institute, Fort Wayne, Indiana
  - Willis Knighton Cancer Center, Shreveport, Louisiana
  - Sandra and Malcolm Berman Cancer Institute, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Renown Regional Medical Center, Reno, Nevada
  - East Carolina University School of Medicine, Greenville, North Carolina
  - The Ohio State University James Cancer Hospital & Solove Research Institute, Columbus, Ohio
  - Ballad Health, Johnson City, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonomi M, Blakaj DM, Kabarriti R, Colvett K, Takiar V, Biagioli M, Bar-Ad V, Goyal S, Muzyka B, Niermann K, Abrouk N, Oronsky B, Reid T, Caroen S, Sonis S, Sher DJ. PREVLAR: Phase 2a Randomized Trial to Assess the Safety and Efficacy of RRx-001 in the Attenuation of Oral Mucositis in Patients Receiving Head and Neck Chemoradiotherapy. Int J Radiat Oncol Biol Phys. 2023 Jul 1;116(3):551-559. doi: 10.1016/j.ijrobp.2022.12.031. Epub 2023 Jan 14. PMID 36646388